CLINICAL TRIAL: NCT03807492
Title: Evaluation and Management for Prostate Oncology, Wellness, and Risk (EMPOWeR)
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Other Study IDs: 18D.644; JT 13180 (Other: JeffTrial Number)
Record Dates: First submitted 2018-12-21; First posted 2019-01-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EMPOWeR Study: This is a cohort study, with initial patient assessments and longitudinal follow-up. Participation of subjects will be indefinite, which will be discussed in the informed consent.

SUMMARY:
The EMPOWeR study is proposed as a cohort study with longitudinal follow-up to determine rates of genetic mutations among men with or at-risk for prostate cancer to address the various facets of genetic education and counseling for optimized genetic assessment and wellness of men. The results will inform practice guidelines and future studies for maximal impact of genetic evaluation of men for inherited prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men with a personal history of prostate cancer
* Unaffected males who are at higher risk for prostate cancer (family history of prostate cancer or African American males)
* Men who previously tested positive for a mutation may be eligible for Specific Aims 2-7
* Men with a known familial mutation
* Men who previously participated in the Genetic Evaluation of Men (GEM) study (IRB#14S.546) will be offered participation in EMPOWeR -

Exclusion Criteria:

* Age < 18 years
* Mental or cognitive impairment that interferes with ability to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As this is a study on prostate cancer, women and children are not included. Minorities meeting eligibility criteria may participate in the study.
Study Population: Any male >18 years with prostate cancer is eligible. Furthermore, unaffected men at higher risk for prostate cancer (family history of prostate cancer or African American males) are also eligible for the study. Men will be approached by their providers or study staff during their clinical appointments for participation. Emails or mailings may also be sent to introduce the study to patients and to contact us for participation. Men who previously participated in the Genetic Evaluation of Men (GEM) study (IRB#14S.546) will be offered participation in EMPOWeR.
Sampling Method: Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Perform genetic testing for men with or at-risk for prostate cancer to determine association of mutations to patient characteristics. | 6 months
  Participants will undergo gene panel testing through a saliva or blood sample. A genetic test summary will be generated to give to participants at disclosure of results. Participants will receive genetic test results in person, by phone or via telehealth. Fisher's exact test will be used to determine association of mutations and variants to patient characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/